CLINICAL TRIAL: NCT07150676
Title: Base de DOnnées Cliniques et Biologiques harmonisées Pour Une REcherche intégrée à la Prise en Charge Des leucémies aiguës Myéloïdes pédiatriques
Brief Title: Harmonized Clinical and Biological Database for Integrated Research Into the Management of Pediatric Acute Myeloid Leukemia
Acronym: DOREMy
Status: Not yet recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP210144
Record Dates: First submitted 2025-08-25; First posted 2025-09-02 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Acute Myeloid Leukemia (AML); Pediatric Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 27 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All children/young adults (<25 years old) with LAM diagnosed in participating French centers
  Interventions: Other: Long term follow-up

INTERVENTIONS:
Other: Long term follow-up — Long term follow-up as part of standard of care

SUMMARY:
The aim of this project is to study the different diagnostic, predictive, and prognostic profiles, as well as their interrelationships (clinical, biological, genetic) in children with Acute Myeloid Leukemia (AML). Despite numerous research projects on separate cohorts, the prognosis for pediatric AML has not improved.

The project therefore consists of pooling research data and existing clinical and biological data from healthcare in a health data warehouse to increase its power.

As these diseases are rare and genetic subgroups even rarer, it is crucial to combine all these data sets into a single database to statistically validate our observations.

The ultimate goal of this project is to reduce the relapse rate and improve the survival rate of pediatric AML by identifying rare, uncharacterized patient subgroups at high risk of relapse, for whom clinical characteristics and outcomes will be compared with omics data, Leukemia Stem Cells signatures, and drug responses to establish accurate and in-depth profiles.

ELIGIBILITY:
All patients under the age of 25 diagnosed with AML in the participating centers in France.

Max Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients already included in a protocol or newly included
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2052-10-01 (Estimated); Study Completion 2052-10-01 (Estimated)

PRIMARY OUTCOMES:
Overall survival | Up to 27 years

SECONDARY OUTCOMES:
Event Free Survival | Up to 27 years
  Event is defined as : relapse, secondary cancer
Cumulative incidence of relapse | Up to 27 years
Cumulative incidence of second cancer | Up to 27 years
Incidence of long-term sequelae | Up to 27 years
  Heart failure, kidney failure, endocrine failure, or any other medical condition covered at 100% by French Social Security

IPD SHARING:
Plan to Share IPD: No